CLINICAL TRIAL: NCT07137429
Title: Platelet Volunteers, Longitudinal and Multi-omic Study
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002298; 002298-H
Record Dates: First submitted 2025-08-21; First posted 2025-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Thrombosis
Keywords: PLATELET FUNCTION; Platelet biology
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Healthy participants, at least 18 years of age

SUMMARY:
Background:

Platelets are a type of blood cell that play a critical role in bleeding, forming blood clots, and healing. Researchers want to know more about platelets work in healthy people. They want to look at how platelets clump together, how blood clots, and how genes and proteins work. They also want to study how these processes change over time and how they are affected by factors such diet, exercise, weight, and new health problems.

Objective:

To study how platelets function in healthy people.

Eligibility:

Healthy people aged 18 years and older.

Design:

Researchers will review participants medical history. They will ask about the participant s family history and any drugs they take.

Participants will have a clinic visit once every 6 or 7 months for 10 years. Each visit will be 2 to 3 hours.

At each visit, participants will have several tests and procedures:

A physical exam, including vital signs. Hip and ankle circumference will be measured.

Urine collection.

Blood tests. About 10 tablespoons of blood will be drawn. Participants will be asked to fast for 10 hours and avoid drugs like aspirin or Advil for 7 days before each draw. Some of the blood may be used for gene studies. Some may be used to create stem cells for research. Stem cells are cells that can be used to make other types of cells.

Surveys and questionnaires. Participants will answer questions about habitual activity, diet, smoking, drugs and alcohol, sleep, illness, and other health issues. These surveys may be done online, via email, or by phone.

DETAILED DESCRIPTION:
Study Description:

This study will serve to provide tissue samples from healthy volunteers for mechanistic studies of platelet function.

Objectives:

Primary Objective: The goal is to obtain blood samples and corresponding derived information to optimize assays, understand variation in these assays due to different sources of variation, and conduct statistical association studies with appropriate designs including cross-sectional analysis, and longitudinal analyses. Environmental variables may include health reports, anthropometric variables, questions on habits and risk factors and medication during the study.

Endpoints:

Primary Endpoints: Establish and validate technical assays and equipment (e.g. platelet aggregation, hemostasis measurements, methylation, RNA-seq, proteomics and WGS, in vitro iPSC generation and bench compound and cellular imaging screening, etc.)

Establish normal physiologic mechanisms and platelet-related parameters in healthy participant samples and how these vary longitudinally and are influenced by variables (e.g., reproducibility, fluctuation with changing diet, exercise, weight and other risk factors or new disease onset)

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures, including fasting at least 10 hours before each blood draw
* Stated willingness to refrain from aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) for 7 days prior to any visits
* Age >= 18 years
* In good general health as evidenced by self-reported medical history

EXCLUSION CRITERIA:

An individual who, by self-report, meets the following criteria will be excluded from participation in this study:

* Current pregnancy or lactation
* Active malignancies known, active known auto-immune disease, known major CVD (e.g., heart attack, stroke, venous thromboembolism, heart failure), severe bleeding history, on regular P2Y12 inhibitors or other antiplatelet treatments for a clinical reason, uncontrolled hypertension or diabetes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy participants, at least 18 years of age
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2041-09-15 (Estimated); Study Completion 2041-09-15 (Estimated)

PRIMARY OUTCOMES:
Establish and validate technical assays and equipment (e.g. platelet aggregation, hemostasis measurements, methylation, RNA-seq, proteomics and WGS, in vitro iPSC. | 10 years
  To provide a mechanism for collection of tissue samples from healthy volunteers for use in research studies relating to platelet biology.The goal is to obtain blood samples and corresponding derived information to optimize assays, understand variation in these assays due to different sources of variation, and conduct statistical association studies with appropriate designs including cross-sectional analysis, and longitudinal analyses. Environmental variables may include health reports, anthropometric variables, questions on habits and risk factors and medication during the study.
Establish normal physiologic mechanisms and platelet-related parameters. How these vary longitudinally and are influenced by variables (e.g., reproducibility, fluctuation with changing diet, exercise, weight and other factors. | 10 years
  To provide a mechanism for collection of tissue samples from healthy volunteers for use in research studies relating to platelet biology.The goal is to obtain blood samples and corresponding derived information to optimize assays, understand variation in these assays due to different sources of variation, and conduct statistical association studies with appropriate designs including cross-sectional analysis, and longitudinal analyses. Environmental variables may include health reports, anthropometric variables, questions on habits and risk factors and medication during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Johnson, Ph.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
See DMSP
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available at the time of associated publication and the duration of availability is expected to be indefinite but will ultimately be determined by the NHLBI.
Access Criteria: Clinical and laboratory data will be collected in the electronic data capture system (CTDB) and analyzed using open-source statistical software packages. Some lab-based research data is collected on specialized instruments and custom processing programs are used to summarize/QC. Those scripts will not be shared unless requested.@@@@@@Data sharing for clinical study (PVLMO)@@@Will be via a separate study accession in dbGaP. Summary level data such as GWAS summary statistics or gene expression level means may be deposited in appropriate public repositories such as NCBI GeoDatasets or the NHLBI GRASP GWAS portal.@@@

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002298-H.html